CLINICAL TRIAL: NCT00571259
Title: Prophylactic Antimicrobial Catheter Lock in Hemodialysis Patients: A Randomized Controlled Clinical Trial
Brief Title: Prophylactic Antimicrobial Catheter Lock
Acronym: ALLOCK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SR001AL
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Bacteremia
Keywords: Sodium citrate; Gentamicin; Prophylaxis; Hemodialysis; Central venous catheter
MeSH Terms: conditions — Bacteremia | interventions — Heparin; Sodium Citrate; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Catheter lock with heparin 1,000 units/mL
  Interventions: Drug: Heparin 1000U/mL
- 2 (Active Comparator): Catheter lock with gentamicin 320 micrograms/mL in sodium citrate 4%
  Interventions: Drug: 4% Sodium Citrate with Gentamicin 320 mcg/mL

INTERVENTIONS:
Drug: Heparin 1000U/mL — A volume sufficient to fill the catheter length will be instilled in both catheter ports post dialysis
  Arms: 1
Drug: 4% Sodium Citrate with Gentamicin 320 mcg/mL — A volume sufficient to fill the catheter length will be instilled in both catheter ports post dialysis
  Arms: 2

SUMMARY:
This is a randomized, double blinded, prospective, multicenter, clinical trial of the use of Heparin versus Gentamicin as a pos-dialysis catheter lock solution.

DETAILED DESCRIPTION:
The study is a randomized, double blinded, prospective, multicenter, clinical trial. All patients requiring vascular access with a tunneled central venous catheter for hemodialysis are eligible for enrollment. Patients will be randomized to receive either Heparin 1,000 U/ml in a volume sufficient to fill the catheter length in both ports or to receive 4% Sodium Citrate with Gentamicin 320 mcg/mL in a volume sufficient to fill the catheter length in both ports.We hypothesize that the device related infection rate in the Citrate/Gentamicin group will be less than the heparin arm.

ELIGIBILITY:
Inclusion Criteria:

* Requires placement of a central venous catheter or currently has a central venous catheter for hemodialysis access.
* Must be at least 18 years old
* Compliant with a dialysis treatment schedule
* Plans to continue hemodialysis treatment and follow-up at the investigational site
* Must be able to care for the exit site independently or have someone who is able to care for the site for them
* Must be able to sign the informed consent document

Exclusion Criteria:

* The subject who has had an infection associated with one or more positive blood cultures is not eligible until 14 days after blood cultures have become negative and clinical resolution of the episode has occurred
* Active exit site or tunnel infection
* Systemic or localized infection that is unresponsive to antibiotic therapy and/or is life threatening
* Known to have antibodies to heparin
* Allergy to pork heparin
* Allergy to gentamicin
* Subject is pregnant
* Known intravenous drug abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2003-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Coplon, MD, Principal Investigator — Satellite Healthcare, Inc.
Locations (1):
- Satellite Healthcare, Inc, Mountain View, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1: Heparin Lock: Dialysis Catheter locked with heparin 1,000 units/mL.
  Heparin 1000U/mL: A volume sufficient to fill the catheter length will be instilled in both catheter ports post dialysis
- 2: Gentamicin Lock: Dialysis Catheter locked with gentamicin 320 micrograms/mL in sodium citrate 4%.
  4% Sodium Citrate with Gentamicin 320 mcg/mL: A volume sufficient to fill the catheter length will be instilled in both catheter ports post dialysis
Period: Overall Study
Arm/Group | 1: Heparin Lock | 2: Gentamicin Lock
Started | 148 | 155
Completed | 4 | 14
Not Completed | 144 | 141

BASELINE CHARACTERISTICS:
Population: All adult patients with either newly placed or existing tunneled cuffed catheters were eligible for enrollment. Patients were excluded if they had an active exit-site or tunnel infection or other systemic or localized infection that was unresponsive to antibiotic therapy and/or was life-threatening. Eligible patients were randomly assigned 1:1 to treatment or control groups.
Groups:
- 1: Heparin Lock: Dialysis catheter locked with heparin 1,000 units/mL post-dialysis.
  Heparin 1000U/mL: A volume sufficient to fill the catheter length will be instilled in both catheter ports post dialysis
- 2: Gentamicin Lock: Dialysis catheter locked with gentamicin 320 micrograms/mL in sodium citrate 4% post-dialysis.
  4% Sodium Citrate with Gentamicin 320 mcg/mL: A volume sufficient to fill the catheter length will be instilled in both catheter ports post dialysis
- Total: Total of all reporting groups
Arm/Group | 1: Heparin Lock | 2: Gentamicin Lock | Total
Number analyzed (Participants) | 148 | 155 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (16.8) | 63.4 (15.6) | 63.1 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 76 | 157
  Male | 67 | 79 | 146
Region of Enrollment [Number; unit: participants]
  United States | 148 | 155 | 303
Diabetes [Count of Participants; unit: Participants] — Percent of subjects in each cohort who were diabetic.
  Participants | 86 | 85 | 171
Dialysis vintage in Months [Median (Full Range); unit: months] — The number of months the subject has been on hemodialysis.
  months | 44.3 [1.1 to 131.8] | 42.4 [0 to 198.5] | 43.32 [0 to 198.5]
Incident Catheters [Count of Participants; unit: Participants] | 15 | 5 | 20
Catheter site [Count of Participants; unit: Participants]
  Internal Jugular | 104 | 113 | 217
  External Jugular | 12 | 12 | 24
  Femoral | 1 | 2 | 3
  Subclavian | 6 | 7 | 13
  Unknown | 25 | 21 | 46

OUTCOME MEASURES:

1. Primary Outcome: Rate of Device-related Bacteremia
Description: Positive blood cultures in a patient whose vascular access is a central venous catheter without another obvious source of infection
Time Frame: 5 years
Population: Episodes of catheter related infections in each group throughout the study.
Measure: Number; unit: Number of infections
Groups:
- 1: Heparin Lock: Dialysis Catheter locked with heparin 1,000 units/mL in a volume sufficient to fill the catheter length and instilled in both catheter ports post-dialysis.
  Heparin 1000U/mL: A volume sufficient to fill the catheter length will be instilled in both catheter ports post dialysis
- 2: Gentamicin Lock: Dialysis Catheter locked with gentamicin 320 micrograms/mL in sodium citrate 4% in a volume sufficient to fill the catheter length and instilled in both catheter ports post-dialysis.
  4% Sodium Citrate with Gentamicin 320 mcg/mL: A volume sufficient to fill the catheter length will be instilled in both catheter ports post dialysis
Arm/Group | 1: Heparin Lock | 2: Gentamicin Lock
Number analyzed (Participants) | 148 | 155
Number of infections | 30 | 11

2. Secondary Outcome: Rate of Catheter Clotting Measured as Requirement for tPA Usage to Maintain Blood Flow
Description: The rate of thrombolytic agent use required to maintain blood flow adequate for dialysis was used as an objective measure of clinically significant catheter clotting.
Time Frame: 5 years
Population: tPA use/1,000 catheter-days
Measure: Number; unit: tPA use/1,000 catheter-days
Groups:
- 1: Heparin Lock: Dialysis Catheter locked with heparin 1,000 units/mL in a volume sufficient to fill the catheter length and instilled in both catheter ports post-dialysis.
- 2: Gentamicin Lock: Dialysis Catheter locked with gentamicin 320 micrograms/mL in sodium citrate 4% in a volume sufficient to fill the catheter length and instilled in both catheter ports post-dialysis.
Arm/Group | 1: Heparin Lock | 2: Gentamicin Lock
Number analyzed (Participants) | 148 | 155
tPA use/1,000 catheter-days | 3.42 | 2.36

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | 1: Heparin Lock | 2: Gentamicin Lock
All-Cause Mortality (participants affected / at risk) | 25/148 | 27/155
Serious Adverse Events (participants affected / at risk) | 25/148 | 27/155
Other Adverse Events (participants affected / at risk) | 0/148 | 0/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Heparin Lock (N=148) | 2: Gentamicin Lock (N=155)
ESRD Related Death (Renal and urinary disorders) | 25 (25) | 27 (27) — Serious adverse events were deaths of dialysis subjects which were related to ESRD or the subject's comorbid conditions, not study related.

LIMITATIONS AND CAVEATS:
The requirement for dialysis facility staff to prepare the treatment intervention prevented a completely blinded study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes